CLINICAL TRIAL: NCT01522716
Title: Mesenchymal Stromal Cells as Treatment of Chronic Graft-versus-host Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New requirements for study approval with the Swedish Medical Products Agency
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Lena von Bahr, Leg läkare, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-cGVH
Record Dates: First submitted 2012-01-24; First posted 2012-02-01 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Graft-Versus-Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal stromal cell treatment (Experimental)
  Interventions: Biological: Mesenchymal stromal cells

INTERVENTIONS:
Biological: Mesenchymal stromal cells — Allogenous mesenchymal stromal cells, to be injected intravenously at a dose of 1-2 million/kg at a frequency of once a month (frequency may be changed during the study if deemed appropriate by investigators) for 6-9 months.

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of mesenchymal stromal cells as treatment for steroid-refractory chronic graft-versus-host disease.

ELIGIBILITY:
Inclusion Criteria:

* Chronic graft-versus-host disease, grade moderate or severe despite at least 3 months treatment with calcineurin inhibitors and steroids OR
* Chronic graft-versus-host disease, grade moderate or severe, where full treatment with calcineurin inhibitors and steroids is impossible due to intolerable side-effects

Exclusion Criteria:

* Active malignancy
* Fulfilling criteria for previously initiated study for treatment of chronic graft-versus-host disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in disease activity according to National Institute of Health criteria | Baseline to 9 months
  Patients are evaluated according to NIH criteria at 3, 6 and (if applicable) 9 months after initialising MSC treatment, and the score compared to baseline score.

SECONDARY OUTCOMES:
Change in disease activity as measured by histological examination | Baseline to 9 months
Change in self-assessed disease activity and quality of life | Baseline to 9 months
Safety (Adverse events, infections and relapse) | 21 months
  Frequency of complications, infections and relapse
Freedom from steroids at 1 year after MSC treatment | 1 year after finishing treatment
  Proportion of patients free from corticosteroids at 1 year after finishing MSC treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Center, Karolinska University Hospital Huddinge, Stockholm, Sweden

REFERENCES:
- [Derived] Boberg E, von Bahr L, Afram G, Lindstrom C, Ljungman P, Heldring N, Petzelbauer P, Garming Legert K, Kadri N, Le Blanc K. Treatment of chronic GvHD with mesenchymal stromal cells induces durable responses: A phase II study. Stem Cells Transl Med. 2020 Oct;9(10):1190-1202. doi: 10.1002/sctm.20-0099. Epub 2020 Jun 23. PMID 32573983